CLINICAL TRIAL: NCT01481129
Title: A Phase 2 Study of MK-2206 in Patients With Relapsed or Refractory Diffuse Large-B Cell Lymphoma
Brief Title: Akt Inhibitor MK2206 in Treating Patients With Relapsed or Refractory Diffuse Large B-Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-00081; NCI-2012-00081 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); LEONB-ET-2011-041; 2011-001970-25; CDR0000716384; ET-2011-041 (Other: Centre Leon Berard); 9022 (Other: CTEP)
Record Dates: First submitted 2011-11-24; First posted 2011-11-29 (Estimated); Results first posted 2017-04-07 (Actual); Last update posted 2017-09-28 (Actual); Status verified 2017-08

CONDITIONS: Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — MK 2206

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Akt inhibitor MK2206) (Experimental): Patients receive Akt inhibitor MK2206 PO once weekly on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Akt Inhibitor MK2206; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study

INTERVENTIONS:
Drug: Akt Inhibitor MK2206 — Given PO
  Other Names: MK2206
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase II trial is studying how well Akt inhibitor MK2206 works in treating patients with relapsed or refractory diffuse large B-cell lymphoma. Akt inhibitor MK2206 may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the antitumor activity of Akt inhibitor MK2206 (MK2206) in terms of objective response rate (ORR) at 4 months (complete response [CR], and partial response [PR]) as per the 2007 International Cheson response criteria.

SECONDARY OBJECTIVES:

I. To evaluate the antitumor activity of MK2206 in terms of ORR at 4 months (CR, unconfirmed complete response [CRu], and PR) as per the 1999 International Cheson response criteria.

II. To determine the duration of response, defined as the time from the date of the best response to the date of progression.

III. To determine the progression-free survival and overall survival of these patients.

IV. To determine the safety of MK2206. V. To identify predictive biomarkers for treatment outcome. (exploratory) VI. To conduct a pharmacodynamic study using FDG-PET scans. (exploratory)

OUTLINE: This a multicenter study.

Patients receive Akt inhibitor MK2206 orally (PO) once weekly on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diffuse large B-cell lymphoma

  * Relapsed or refractory disease
* Measurable disease

  * At least one measurable lymph node mass that is > 1.5 cm in two perpendicular dimensions and that has not been previously irradiated or has grown since previous irradiation

    * Dominant lymph node masses include up to 6 nodal masses that are clearly measurable in 2 perpendicular dimensions and > 1.5 cm in each dimension
    * Measurement may be by radiographic imaging
    * If there are lymph node masses in the mediastinum or pelvis larger than 1.5 cm in 2 perpendicular dimensions, they should always be chosen as dominant masses
    * The dominant masses should be from as disparate regions of the body as possible
  * Measurable sites of disease are also extra-nodal sites such as splenic nodules and hepatic nodules that are thought to contain lymphoma, and are greater than 1 cm in the longest transverse dimension
* Must have received at least two prior treatment lines; there is no maximal limit on the number of prior therapies

  * Prior treatment must include CHOP (cyclophosphamide, doxorubicin, vincristine, and prednisolone)-like chemotherapy in combination with rituximab

    * Rituximab used alone is not considered as a separate regimen
    * Salvage treatment, mobilization chemotherapy, high-dose chemotherapy, and planned post-transplant therapy should be considered as one regimen
  * Relapsed or refractory patients who are candidates for high-dose chemotherapy and autologous or allogeneic stem cell transplantation are not eligible
* Tumor tissue sample must be available for pathological review
* No known CNS involvement
* ECOG performance status < 2 (Karnofsky > 60%)
* Life expectancy > 4 months
* Absolute neutrophil count >= 1,500/µL
* Platelets >= 100,000/µL (>= 75,000/µL if the bone marrow is involved)
* Total bilirubin =< 1.5 X institutional upper limit of normal (ULN)
* AST(SGOT)/ALT(SGPT) =< 2.5 X ULN
* Calculated creatinine clearance >= 50 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Women of child-bearing potential and men must agree to use adequate contraception
* Must be able to swallow whole tablets

  * Nasogastric or G-tube administration is not allowed
  * Tablets must not be crushed or chewed
* Patients with French Social Security in compliance with the French law relating to biomedical research allowed
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to MK2206 tablets
* Hyperglycemia should be well controlled on oral agents
* Cardiovascular baseline QTcF =< 450 msec (male) or QTcF =< 470 msec (female)
* No uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* No HIV-positive patients on combination antiretroviral therapy
* No patients with malabsorption syndrome or other condition that would interfere with intestinal absorption
* No patients with clinically important history of liver disease, including viral or other hepatitis or cirrhosis
* No prior history of malignancies other than lymphoma (except for basal cell or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or breast) unless the subject has been free of the disease for >= 3 years
* Must have recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients must have discontinued all prior therapies for at least 5 times the half-life of all prior anticancer therapies before study entry
* Prior treatment could include high-dose chemotherapy with autologous stem-cell transplantation if patients had progressed >= 3 months after this treatment
* No chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C)
* Patients must not be receiving any other investigational agents
* No other investigational or commercial agents or therapies may be administered with the intent to treat the patient's malignancy
* No concurrent radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2011-12 (Actual); Primary Completion 2013-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herve Ghesquieres, Principal Investigator — Centre Leon Berard
Locations (9):
- France (9):
  - Hopitaux de Paris, Vellefaux, Paris
  - Institut Bergonie Cancer Center, Bordeaux
  - Henri Mondor University-Hospital Center, Créteil
  - Hospital Claude Huriez Chru, Lille
  - Centre Leon Berard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Hopital Saint Louis, Paris
  - Centre Hospitalier Lyon-Sud, Pierre-Bénite
  - Institut Gustave Roussy, Villejuif

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Akt Inhibitor MK2206)
Started | 22
Completed | 22
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Akt Inhibitor MK2206)
Number analyzed (Participants) | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 10
Age, Continuous [Mean (Full Range); unit: years] | 64.9 [43.7 to 85.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 12
Region of Enrollment [Number; unit: participants]
  France | 22

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate According to the International Response Criteria for DLBCL (Cheson 2007)
Description: Rate of CR + PR according to Cheson 2007 after 4 months of treatment
Time Frame: Up to 4 months
Measure: Number; unit: objective response
Arm/Group | Treatment (Akt Inhibitor MK2206)
Number analyzed (Participants) | 22
objective response | 0

2. Secondary Outcome: Duration of Response
Description: Described in responding subjects using descriptive statistics (median, extreme values, etc.).
Time Frame: up to 4 years
Population: No responses were observed
Arm/Group | Treatment (Akt Inhibitor MK2206)
Number analyzed (Participants) | 0

3. Secondary Outcome: Overall Survival
Description: Analyzed using the Kaplan-Meier method. The median survival rates will be reported with a 95% confidence interval. Median follow-up will be calculated using the reverse Kaplan-Meier method.
Time Frame: From the date of inclusion to the date of death from any cause, assessed up to 4 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Akt Inhibitor MK2206)
Number analyzed (Participants) | 22
months | 9.6 [2.8 to 18.8]

4. Secondary Outcome: Progression-free Survival (PFS)
Description: as for outcome 3
Time Frame: From the date of inclusion to the date of first documented disease progression, relapse or death from any cause, assessed up to 4 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Akt Inhibitor MK2206)
Number analyzed (Participants) | 22
months | 1.71 [0.8 to 1.8]

5. Secondary Outcome: Toxicity as Assessed by Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0
Time Frame: Up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Akt Inhibitor MK2206)
Number analyzed (Participants) | 19
Participants | 19

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Treatment (Akt Inhibitor MK2206)
Serious Adverse Events (participants affected / at risk) | 8/19
Other Adverse Events (participants affected / at risk) | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Akt Inhibitor MK2206) (N=19)
vomiting (Gastrointestinal disorders) | 1
diarrhea (Gastrointestinal disorders) | 1
Gastro intestinal bleeding (Gastrointestinal disorders) | 1
Hyperglycemia (Endocrine disorders) | 1
Drug overdose accidental (Injury, poisoning and procedural complications) | 1
Pericarditis (Cardiac disorders) | 1
Pulmonary embolism (Vascular disorders) | 1
Arrhythmia supraventricular (Cardiac disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Drug allergy (Immune system disorders) | 1
General physical health deterioration (General disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Distress respiratory (Respiratory, thoracic and mediastinal disorders) | 1
Hemolytic uremic syndrome (Blood and lymphatic system disorders) | 1
Death (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Akt Inhibitor MK2206) (N=19)
arythmia (Cardiac disorders) | 1
heart palpitations (Cardiac disorders) | 1
tachycardia (Cardiac disorders) | 1
mouth ulcers (Skin and subcutaneous tissue disorders) | 1
cutaneous eruption (Skin and subcutaneous tissue disorders) | 3
cutaneous erythema (Skin and subcutaneous tissue disorders) | 1
papule (Skin and subcutaneous tissue disorders) | 1
prurigo (Skin and subcutaneous tissue disorders) | 1
prurit (Skin and subcutaneous tissue disorders) | 1
cutaneous rash (Skin and subcutaneous tissue disorders) | 1
maculopapular rash (Skin and subcutaneous tissue disorders) | 3
toxidermia (Skin and subcutaneous tissue disorders) | 1
dysgueusia (Nervous system disorders) | 1
encephalopathy (Nervous system disorders) | 1
paresthesia (Nervous system disorders) | 1
diarrhea (Gastrointestinal disorders) | 4
digestive bleeding (Gastrointestinal disorders) | 1
nausea (Gastrointestinal disorders) | 4
stomatitis (Gastrointestinal disorders) | 1
vomiting (Gastrointestinal disorders) | 2
uremic hemolytic syndrome (Blood and lymphatic system disorders) | 1
epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
hypertension (Cardiac disorders) | 2
hypotension (Cardiac disorders) | 1
thrombosis (Cardiac disorders) | 1
increase bilrubin (Investigations) | 1
creatinine clearance decrease (Investigations) | 2
creatinine increase (Investigations) | 1
eosinophil increase (Investigations) | 1
GGT increase (Investigations) | 2
anemia (Investigations) | 2
QT prolongation (Investigations) | 2
leucopenia (Investigations) | 3
lymphopenia (Investigations) | 3
neutrophil decrease (Investigations) | 5
alkaline phosphatase increase (Investigations) | 1
thrombopenia (Investigations) | 5
SGOT increase (Investigations) | 1
albumine decrease (Metabolism and nutrition disorders) | 1
calcium decrease (Metabolism and nutrition disorders) | 1
glycaemia increase (Metabolism and nutrition disorders) | 6
appetite loss (Metabolism and nutrition disorders) | 1
decreases phosphorus (Metabolism and nutrition disorders) | 4
asthenia (General disorders) | 4
chest pain (General disorders) | 1
fatigue (General disorders) | 3
lower limbs oedema (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less